CLINICAL TRIAL: NCT03485794
Title: Metabolic Profiling of Peripheral Blood Mononuclear Cells (PBMCs) by LC-MS in Prostate Cancer Patients
Brief Title: Collection of Blood in Studying Metabolites in Patients With Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4P-17-8; NCI-2017-02078 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-17-8 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, PBMCs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (biospecimen collection): Patients undergo collection of blood for metabolic profiling via LC/Q-TOF/MS.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot research trial utilizes the collection of blood in studying metabolites in patients with prostate cancer. Metabolites are the small molecule products of cellular metabolism that are produced naturally in all living cells. Collecting blood in order to study metabolites may help doctors monitor and treat prostate cancer more effectively.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop blood sample collection and preparation procedures for reliable, meaningful metabolomic profiling of peripheral blood mononuclear cells (PBMCs) by liquid chromatography/quadruple-time of flight/mass spectrometry (LC/Q-TOF/MS) that can be implemented in a clinical setting.

II. Optimize data analysis methods and software usage to create a metabolic profile for patients at the time of blood collection.

III. Compare metabolite profiles of isolated PBMCs versus (vs.) other blood fractions (plasma, red blood cells [RBCs], and whole blood).

IV. Identify elements of the PBMC metabolite profile that may correlate to patient disease state.

OUTLINE:

Patients undergo collection of blood for metabolic profiling via LC/Q-TOF/MS.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have histologically confirmed prostate cancer
* Provide written consent/authorization to participate in this study
* Have no signs or symptoms of active infection
* Exhibit a willingness to comply with the experimental procedures as outlined in this protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer who are patients at the University of Southern California (USC) Westside Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Blood sample collection | Baseline
  The blood will be used to analyze the metabolites produced by white blood cells.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Katz, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States